CLINICAL TRIAL: NCT00091962
Title: Treatment of Depression Following Bypass Surgery
Brief Title: Effectiveness of Depression Treatment Following Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Bruce Rollman, Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 164; R01HL070000 (NIH)
Record Dates: First submitted 2004-09-20; First posted 2004-09-23 (Estimated); Results first posted 2016-04-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-03

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Depression | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Depressed Intervention (Experimental): Telephone-based, nurse-delivered Collaborative Care program for depression; Involving: Psychoeducation; workbook for depression self-care; initiation or adjustment of antidepressant pharmacotherapy prescribed under their PCPs' direction; referral to mental health specialist
  Interventions: Behavioral: Psychoeducation; Treatment recommendations; Drug: Pharmacotherapy
- Depressed Usual Care (Active Comparator): "Usual care" for depression; feedback of the depression finding by the study team
  Interventions: Other: Usual Care
- Non-Depressed Control Group (No Intervention): Non-depressed control group

INTERVENTIONS:
Behavioral: Psychoeducation; Treatment recommendations — Counseling program
  Arms: Depressed Intervention
Drug: Pharmacotherapy — Recommendations to patients' PCP for medication to treat depression
  Arms: Depressed Intervention
Other: Usual Care — Physicians' Usual care
  Arms: Depressed Usual Care

SUMMARY:
The purpose of this study is to treat depression in patients who have undergone coronary artery bypass graft (CABG).

DETAILED DESCRIPTION:
BACKGROUND:

Cardiovascular disease morbidity and mortality is an important health issue. Depression has emerged as a risk factor for increased morbidity and mortality in patients with coronary heart disease. CABG is a surgical procedure that is specifically directed to improvement in quality of life for patients with severe coronary artery disease, though its impact on mortality is questionable. Patients with depression after CABG are found to not demonstrate sufficient improvement in quality of life, resulting in a significantly higher level of healthcare costs.

DESIGN NARRATIVE:

In this randomized study, 300 patients who show elevated levels of depressive symptoms at 3 to 5 days following CABG and at 2 weeks after hospital discharge will be recruited. They will be randomized to receive either 1) their physician's "usual care" for depression, or 2) a stepped collaborative care program involving a telephone-based nurse care manager. The nurse care manager will contact patients at regular intervals to assess treatment preferences for depression (e.g., counseling, self-management workbook, pharmacotherapy, or specialty referral), promote adherence with care, and monitor the therapeutic response in concert with patient's primary care physicians and under the supervision of a study clinician. One hundred and fifty nondepressed post-CABG patients will be randomly selected to serve as a control cohort to facilitate comparisons with the depressed patients on various baseline and follow-up measures, and to better understand the benefits derived from depression treatment (total N=450). Blinded telephone assessments will be conducted at 2, 4, 8, and 12 months post CABG and then every 6 months until the last patient completes his/her 8-month assessment (range: 8-44 months follow-up). Intent-to-treat analyses will be used to test the primary hypothesis that the intervention will produce at least a clinically meaningful 0.5 effect size improvement in health related quality of life (HRQoL) at 8 months post CABG, as measured by the SF-36 Mental Component Summary score, compared to patients who receive their primary care physician's "usual care" for depression. The secondary hypotheses are that compared to "usual care" patients, intervention patients will 1) experience higher levels of functional status, and lower levels of depressive symptoms, risk for future cardiovascular events, and health services costs, and 2) report similar levels of HRQoL as nondepressed post-CABG patients. Providing evidence-based, stepped, collaborative care treatment for post-CABG depression may be an ideal method for organized health care delivery systems to improve outcomes. The focus on HRQoL and health services costs will facilitate comparisons of the benefits derived from the intervention to that of other established treatments of cardiovascular risk factors and care for other chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Recently underwent CABG (combined or redo procedure) at one of 8 Pittsburgh area study hospitals
* A PHQ score greater than 10 OR if nondepressed control, a PHQ score less than 5 at both 2 days post CABG to the date of discharge following CABG and when reassessed 2 weeks after hospital discharge
* Folstein Mini-Mental State Examination (MMSE) score greater than or equal to 24
* Able to be evaluated and treated for depression as an outpatient post CABG
* Has a household telephone

Exclusion Criteria:

* Presently in treatment with a mental health specialist
* Actively suicidal
* History of psychotic illness
* History of bipolar illness according to subject self-report and past medical history
* Current alcohol dependence or other substance abuse as evidenced by chart review and the CAGE questionnaire
* Organic mood syndromes, including those secondary to medical illness or drugs
* Presence of non-cardiovascular conditions that are likely to be fatal within 1 year
* Unstable medical condition as indicated by history, physical, and/or laboratory findings
* Previous enrollment in the study cohort
* Non-English speaking, illiterate, or possessing any other communication barrier
* If nondepressed control, current or previous diagnosis or treatment of depression

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2003-08; Primary Completion 2008-06 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce L. Rollman, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Rollman BL, Belnap BH, LeMenager MS, Mazumdar S, Schulberg HC, Reynolds CF 3rd. The Bypassing the Blues treatment protocol: stepped collaborative care for treating post-CABG depression. Psychosom Med. 2009 Feb;71(2):217-30. doi: 10.1097/PSY.0b013e3181970c1c. Epub 2009 Feb 2. PMID 19188529
- [Result] Morone NE, Weiner DK, Belnap BH, Karp JF, Mazumdar S, Houck PR, He F, Rollman BL. The impact of pain and depression on recovery after coronary artery bypass grafting. Psychosom Med. 2010 Sep;72(7):620-5. doi: 10.1097/PSY.0b013e3181e6df90. Epub 2010 Jun 18. PMID 20562371
- [Result] Rollman BL, Belnap BH, LeMenager MS, Mazumdar S, Houck PR, Counihan PJ, Kapoor WN, Schulberg HC, Reynolds CF 3rd. Telephone-delivered collaborative care for treating post-CABG depression: a randomized controlled trial. JAMA. 2009 Nov 18;302(19):2095-103. doi: 10.1001/jama.2009.1670. Epub 2009 Nov 16. PMID 19918088
- [Result] Tindle H, Belnap BH, Houck PR, Mazumdar S, Scheier MF, Matthews KA, He F, Rollman BL. Optimism, response to treatment of depression, and rehospitalization after coronary artery bypass graft surgery. Psychosom Med. 2012 Feb-Mar;74(2):200-7. doi: 10.1097/PSY.0b013e318244903f. Epub 2012 Jan 27. PMID 22286847
- [Result] Ghesquiere A, Shear MK, Gesi C, Kahler J, Belnap BH, Mazumdar S, He F, Rollman BL. Prevalence and correlates of complicated grief in adults who have undergone a coronary artery bypass graft. J Affect Disord. 2012 Feb;136(3):381-5. doi: 10.1016/j.jad.2011.11.018. Epub 2011 Dec 29. PMID 22209126
- [Result] Rollman BL, Belnap BH. The Bypassing the Blues trial: collaborative care for post-CABG depression and implications for future research. Cleve Clin J Med. 2011 Aug;78 Suppl 1:S4-12. doi: 10.3949/ccjm.78.s1.01. PMID 21972329
- [Result] Schulberg HC, Belnap BH, Houck PR, Mazumdar S, Reynolds CF 3rd, Rollman BL. Treating post-CABG depression with telephone-delivered collaborative care: does patient age affect treatment and outcome? Am J Geriatr Psychiatry. 2011 Oct;19(10):871-80. doi: 10.1097/JGP.0b013e31820d9416. PMID 21946803
- [Result] Donohue JM, Belnap BH, Men A, He F, Roberts MS, Schulberg HC, Reynolds CF 3rd, Rollman BL. Twelve-month cost-effectiveness of telephone-delivered collaborative care for treating depression following CABG surgery: a randomized controlled trial. Gen Hosp Psychiatry. 2014 Sep-Oct;36(5):453-9. doi: 10.1016/j.genhosppsych.2014.05.012. Epub 2014 May 21. PMID 24973911
- [Result] Meyer T, Belnap BH, Herrmann-Lingen C, He F, Mazumdar S, Rollman BL. Benefits of collaborative care for post-CABG depression are not related to adjustments in antidepressant pharmacotherapy. J Psychosom Res. 2014 Jan;76(1):28-33. doi: 10.1016/j.jpsychores.2013.10.017. Epub 2013 Nov 5. PMID 24360138
- [Result] Morone NE, Belnap BH, He F, Mazumdar S, Weiner DK, Rollman BL. Pain adversely affects outcomes to a collaborative care intervention for anxiety in primary care. J Gen Intern Med. 2013 Jan;28(1):58-66. doi: 10.1007/s11606-012-2186-2. Epub 2012 Aug 10. PMID 22878857
- [Result] Herbeck Belnap B, Schulberg HC, He F, Mazumdar S, Reynolds CF 3rd, Rollman BL. Electronic protocol for suicide risk management in research participants. J Psychosom Res. 2015 Apr;78(4):340-5. doi: 10.1016/j.jpsychores.2014.12.012. Epub 2014 Dec 27. PMID 25592159
- [Derived] Waterman LA, Belnap BH, Gebara MA, Huang Y, Abebe KZ, Rollman BL, Karp JF. Bypassing the blues: Insomnia in the depressed post-CABG population. Ann Clin Psychiatry. 2020 Feb;32(1):17-26. PMID 31675390

RESULTS

PARTICIPANT FLOW:
Groups:
- Depressed Intervention: Collaborative care program for depression involving a telephone-based nurse care manager
  Counseling: Counseling program
  Pharmacotherapy: Medication to treat depression
- Depressed Usual Care: Control group will receive usual care for depression
  Usual Care: Usual care for depression
Period: Overall Study
Arm/Group | Depressed Intervention | Depressed Usual Care | Non-Depressed Control Group
Started | 150 | 152 | 151
Completed | 150 | 152 | 151
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-Depressed Control: Observational only
- Total: Total of all reporting groups
Arm/Group | Depressed Intervention | Depressed Usual Care | Non-Depressed Control | Total
Number analyzed (Participants) | 150 | 152 | 151 | 453
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 85 | 84 | 60 | 229
  >=65 years | 65 | 68 | 91 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10.8) | 64 (11.2) | 66 (9.6) | 65 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 56 | 56 | 181
  Male | 81 | 96 | 95 | 272
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 2 | 5
  Not Hispanic or Latino | 147 | 152 | 149 | 448
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 17 | 10 | 25 | 52
  White | 132 | 142 | 122 | 396
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 150 | 152 | 151 | 453

OUTCOME MEASURES:

1. Primary Outcome: Generic Mental Health-Related Quality of Life
Description: The 36-item Medical Outcomes Study Form (v.2) Mental Component Scale (SF-36 MCS). Range 0-100; Population norm is 50 with standard deviation of 10. Higher scores are better.
  Ware J, Kosinski M, Keller S. SF-36 Physical and Mental Health Summary Scales: A User's Manual. 2nd ed. Boston, MA: New England Medical Center; 1994.
Time Frame: Measured 8 months post-CABG
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Depressed Intervention: Telephone-based, nurse-delivered Collaborative Care program for depression; Involving: Psychoeducation; workbook for depression self-care; initiation or adjustment of antidepressant pharmacotherapy prescribed under their PCPs' direction; referral to mental health specialist
  Psychoeducation; Treatment recommendations: Counseling program
  Pharmacotherapy: Medication to treat depression
- Depressed Usual Care: "Usual care" for depression by patients' PCP
- Non-Depressed Control: Non-depressed control group with no intervention
Arm/Group | Depressed Intervention | Depressed Usual Care | Non-Depressed Control
Number analyzed (Participants) | 150 | 152 | 151
units on a scale | 50.0 (1.0) | 46.2 (1.1) | 57.2 (0.5)

2. Secondary Outcome: Hamilton Rating Scale for Depression
Description: The 17-item Depression Interview and Structured Hamilton (DISH) version of the Hamilton Rating Scale for Depression Standard provides an accurate DSM-IV diagnosis of a cardiac patient's mood disorder and a reliable HRS-D score. Range 0-52. Higher scores are worse. Psychosom Med. 2002;64(6):897-905
Time Frame: 8 months post CABG
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Non-Depressed Control Group: Non-depressed groups as Control to see the natural course of recovery after CABG
Arm/Group | Depressed Intervention | Depressed Usual Care | Non-Depressed Control Group
Number analyzed (Participants) | 150 | 152 | 151
units on a scale | 9.0 (0.7) | 11.4 (0.7) | 3.8 (0.3)
Statistical Analysis 1: Comparison: Depressed Intervention vs Depressed Usual Care; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — repeated measures mixed-effect model with treatment, time (4 time points), and sex; all 2- and 3-factor interaction terms with subject intercepts were treated as a random effect to account for individual differences at randomization; Mean Difference (Final Values) = 0.001

3. Secondary Outcome: Generic Physical Health-Related Quality of Life
Description: The 36-item Medical Outcomes Study Form (v.2) Physical Component Scale (SF-36 PCS). Range 0-100; Population norm is 50 with standard deviation of 10. Higher scores are better.
  Ware J, Kosinski M, Keller S. SF-36 Physical and Mental Health Summary Scales: A User's Manual. 2nd ed. Boston, MA: New England Medical Center; 1994.
Time Frame: 8 months post CABG
Measure: Mean (Standard Error); unit: participants
Arm/Group | Depressed Intervention | Depressed Usual Care | Non-Depressed Control
Number analyzed (Participants) | 150 | 152 | 151
participants | 44.0 (0.8) | 41.4 (0.8) | 48.7 (0.7)

4. Secondary Outcome: Disease-Specific Health-Related Quality of Life
Description: The 12-item Duke Activity Status Index (DASI). Scores range from 0-58.2, and higher scores the better the functional capacity (Am J Cardiol. 1989;64(10):651-654).
Time Frame: 8 months post CABG
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Depressed Intervention | Depressed Usual Care | Non-Depressed Control
Number analyzed (Participants) | 150 | 152 | 151
units on a scale | 25.2 (1.0) | 21.4 (1.0) | 33.2 (1.1)

ADVERSE EVENTS:
Arm/Group | Depressed Intervention | Depressed Usual Care | Non-Depressed Control
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/152 | 0/151
Other Adverse Events (participants affected / at risk) | 0/150 | 0/152 | 0/151

LIMITATIONS AND CAVEATS:
Selection bias if patients with severe depression were less likely to participate in our screening procedure. Also, the trial recruited just from one U.S. region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No